CLINICAL TRIAL: NCT00241241
Title: Multicenter Phase 2 Study of Efficacy and Safety of Pegylated Interferon-alfa 2a in Polycythemia Vera Patients
Brief Title: Efficacy and Safety of Pegylated Interferon Alfa in Polycythemia Vera
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PV-Nord (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVN1
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Polycythemia Vera
Keywords: myeloproliferative disorder; polycythemia vera; interferon
MeSH Terms: conditions — Polycythemia Vera; Myeloproliferative Disorders | interventions — peginterferon alfa-2a

INTERVENTIONS:
Drug: pegylated interferon-alfa 2a

SUMMARY:
Interferon alfa is an effective treatment of polycythemia vera (PV), but about 20% of patients discontinue their treatment because of side effects and treatment schedule (three times per week administration). The pegylated form of interferon alfa-2a has shown a better tolerance in hepatitis patients and is administered only once a week. The purpose of this study is to determine efficacy and safety of pegylated interferon alfa-2a in the treatment of PV patients.

DETAILED DESCRIPTION:
The aim of PV treatment is to reduce the risk of vascular thrombosis without enhancing the long-term risk of evolution toward myelofibrosis or MDS/AL. Although currently controversial, phlebotomies have been shown in the old PVSG01 study to increase the risk of both thrombosis and myelofibrosis. On the other hand, currently available cytoreductive treatments have been shown to efficiently reduce the thrombotic risk, but were demonstrated (32P, busulfan, chlorambucil) or suspected (pipobroman, hydroxyurea) to enhance the risk of evolution to MDS/AL. In fact, the main widely used cytoreductive treatment, when indicated, is hydroxyurea (HU). This drug is very efficient to control myeloproliferation with a response rate of 80 to 90%. It is generally well tolerated, even if long term toxicity leads to treatment change in 10% of cases. Although no prospective study has yet clearly demonstrated its leukemogenic potential in PV, a non-leukemogenic alternative treatment is highly warranted, especially for younger patient.

Interferon (IFN) alpha is a promising agent in PV both because of good efficacy and absence of leukemogenic risk. Expanded experience with IFN-alpha was recently reported, showing a control of erythrocytosis in approximately 75% of patients. A similar percentage of patients also have resolution of disease-related symptoms, in particular a reduction in spleen size and relief from intractable pruritus. In some cases, long-term persisting remissions after treatment discontinuation have been observed as well as demonstration of eradication of the myeloproliferative clone. However, 20% of patients may not tolerate the treatment because of side effects. Furthermore, the treatment schedule (three times per week administration) may be a factor reducing long-term compliance to this drug.

In this regard, pegylated-IFN could be a major drug in PV. The weekly administration and better tolerance by comparison to IFN reported in hepatitis patients could allow to obtain results similar to chemotherapy in terms of compliance to treatment and efficacy, with a major advantage, its lack of mutagenicity.

ELIGIBILITY:
Inclusion Criteria:

* polycythemia vera diagnosed according to PVSG criteria, modified by Pearson
* Previously untreated patients or patients treated by phlebotomy only or HU or pipobroman for less than 2 years
* Age 18 to 65 years
* Signed informed consent

Exclusion Criteria:

* Contra indication for interferon
* Severe renal or liver disease
* ECOG performance status > 2
* Pregnancy
* Uncontrolled endocrine disorders except well regulated hyperthyroidism and diabetes
* Severe concomitant heart failure or psychiatric disorder
* Patients receiving an other investigational treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-09; Primary Completion 2006-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
response rate after one year of treatment

SECONDARY OUTCOMES:
safety
molecular response

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Kiladjian, MD, Principal Investigator — PV-Nord; Pierre Fenaux, MD, PhD, Study Chair — PV-Nord; Christine Chomienne, MD, PhD, Study Chair — PV-Nord; Sylvia Bellucci, MD, Study Chair — PV-Nord; Bruno Cassinat, MD, Study Chair — PV-Nord; Marie-Jose Grange, MD, Study Chair — PV-Nord; Nathalie Cambier, MD, Study Chair — PV-Nord; Jean-Francois Bernard, MD, Study Chair — PV-Nord; Philippe Rousselot, MD, Study Chair — PV-Nord
Locations (5):
- France (5):
  - Hopital Avicenne, Bobigny
  - Hopital Huriez, Lille
  - Hopital Dupuytren, Limoges
  - Hopital Lariboisiere, Paris
  - Hopital Saint-Louis, Paris

REFERENCES:
- [Background] Berk PD, Goldberg JD, Donovan PB, Fruchtman SM, Berlin NI, Wasserman LR. Therapeutic recommendations in polycythemia vera based on Polycythemia Vera Study Group protocols. Semin Hematol. 1986 Apr;23(2):132-43. PMID 3704665
- [Background] Fruchtman SM, Mack K, Kaplan ME, Peterson P, Berk PD, Wasserman LR. From efficacy to safety: a Polycythemia Vera Study group report on hydroxyurea in patients with polycythemia vera. Semin Hematol. 1997 Jan;34(1):17-23. No abstract available. PMID 9025158
- [Background] Kiladjian JJ, Bernard JF, Fenaux P. Is life expectancy of polycythemia vera patients clearly different from that of the general population? Am J Med. 2005 May;118(5):565; author reply 565-6. doi: 10.1016/j.amjmed.2004.12.026. No abstract available. PMID 15866263
- [Background] Lengfelder E, Berger U, Hehlmann R. Interferon alpha in the treatment of polycythemia vera. Ann Hematol. 2000 Mar;79(3):103-9. doi: 10.1007/s002770050563. PMID 10803930
- [Background] Streiff MB, Smith B, Spivak JL. The diagnosis and management of polycythemia vera in the era since the Polycythemia Vera Study Group: a survey of American Society of Hematology members' practice patterns. Blood. 2002 Feb 15;99(4):1144-9. doi: 10.1182/blood.v99.4.1144. PMID 11830459
- [Derived] Kiladjian JJ, Cassinat B, Chevret S, Turlure P, Cambier N, Roussel M, Bellucci S, Grandchamp B, Chomienne C, Fenaux P. Pegylated interferon-alfa-2a induces complete hematologic and molecular responses with low toxicity in polycythemia vera. Blood. 2008 Oct 15;112(8):3065-72. doi: 10.1182/blood-2008-03-143537. Epub 2008 Jul 23. PMID 18650451
- [Derived] Kiladjian JJ, Cassinat B, Turlure P, Cambier N, Roussel M, Bellucci S, Menot ML, Massonnet G, Dutel JL, Ghomari K, Rousselot P, Grange MJ, Chait Y, Vainchenker W, Parquet N, Abdelkader-Aljassem L, Bernard JF, Rain JD, Chevret S, Chomienne C, Fenaux P. High molecular response rate of polycythemia vera patients treated with pegylated interferon alpha-2a. Blood. 2006 Sep 15;108(6):2037-40. doi: 10.1182/blood-2006-03-009860. Epub 2006 May 18. PMID 16709929